CLINICAL TRIAL: NCT03958955
Title: Efficacy and Safety of Twice-daily Application of Delgocitinib Cream 20 mg/g for 6 Weeks in Subjects With Active Discoid Lupus Erythematosus.
Brief Title: Efficacy and Safety of Delgocitinib Cream in Discoid Lupus Erythematosus.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to recruitment challenges.
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXP-1373; 2018-003615-22 (EudraCT Number)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Results first posted 2021-06-28 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2020-05

CONDITIONS: Discoid Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Discoid

STUDY DESIGN:
Intervention Model Description: This was a phase 2a, within-subject trial design, where all subjects were treated with active treatment on one DLE target lesion and vehicle treatment on another DLE target lesion.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Delgocitinib cream 20 mg/g (Experimental): Delgocitinib cream applied twice daily for 6 weeks
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream vehicle (Placebo Comparator): Delgocitinib cream vehicle applied twice daily for 6 weeks
  Interventions: Drug: Delgocitinib cream vehicle

INTERVENTIONS:
Drug: Delgocitinib cream — Cream for topical application.
  Other Names: LEO 124249 cream
  Arms: Delgocitinib cream 20 mg/g
Drug: Delgocitinib cream vehicle — The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
  Other Names: LEO 124249 cream vehicle
  Arms: Delgocitinib cream vehicle

SUMMARY:
This was a double-blind, multi-centre, randomised, vehicle-controlled, within-subject phase 2a trial. The trial was designed to establish the efficacy and safety of delgocitinib cream in the treatment of adult subjects with discoid lupus erythematosus (DLE).

ELIGIBILITY:
Main Inclusion Criteria:

* Histopathological findings (current or previous) consistent with clinical diagnosis of DLE.
* Unequivocal clinical diagnosis of 2 active DLE target lesions that were <6 months old and amenable for clinical evaluation. This included lesions located on the scalp if they fulfilled all lesion-specific eligibility criteria.
* Target lesion IGA score of at least moderate severity (≥3) at screening and baseline.
* Target lesion erythema score ≥2 at screening and baseline.

Main Exclusion Criteria:

* Target lesion dyspigmentation score of 2 at screening or baseline.
* Target lesion scarring/atrophy score of 2 at screening or baseline.
* Target lesion scarring alopecia score of >0 in scalp lesions at screening or baseline.
* Medical history of systemic lupus erythematosus (SLE) with clinically significant organ involvement (American College of Rheumatology SLE classification criteria no. 6 to 9) including SLE-related pleuritis or pericarditis (by clinical evaluation and electrocardiogram), and neurologic, renal, and/or other major SLE-related organ system involvement. SLE joint involvement was acceptable.
* Subjects with unstable or significant SLE disease activity findings that would, by its progressive nature and/or severity, interfere with the trial evaluation, completion, and/or procedures per the investigator's discretion.
* Other skin conditions at screening or baseline that would interfere with the evaluation of DLE.
* Immunosuppressive/immunomodulating therapy with e.g. methotrexate, cyclosporine, azathioprine, retinoids (both topical and systemic), or dapsone within 4 weeks prior to baseline.
* Systemic prednisolone >7.5 mg/day or changed dose within 4 weeks prior to baseline (nasal and inhaled corticosteroids were allowed).
* Treatment with the following medications:

  * Oral antimalarial treatment with hydroxychloroquine >6.5 mg/kg body weight/day, or chloroquine >4 mg/kg body weight/day, or changed dose within 12 weeks prior to baseline.
  * Quinacrine combined with either hydroxychloroquine or chloroquine within 12 weeks prior to baseline.
  * Drugs known to interact with antimalarials (e.g. digoxin, cimetidine) within 12 weeks prior to baseline.
* Treatment with topical corticosteroids, calcineurin inhibitors, and phosphodiesterase-4 (PDE-4) inhibitors within 2 weeks prior to baseline.
* Use of systemic antibiotics or cutaneously applied antibiotics on the target lesions within 2 weeks prior to baseline.
* Ultraviolet (UV) therapy within 2 weeks prior to baseline.
* Any procedure impairing the skin barrier (e.g. incision) within 2 cm from the border of any of the target lesions within 4 weeks prior to baseline.
* Receipt of live (attenuated) vaccines within 4 weeks prior to baseline.
* Treatment with any marketed biological therapy or investigational biologic agents:

  * Any cell-depleting agents including but not limited to rituximab: within 6 months prior to baseline, or until lymphocyte count returned to normal, whichever was longer.
  * Other biologics: within 3 months or 5 half-lives, whichever was longer, prior to baseline.
* Unstable or fluctuating use of tobacco within 1 month prior to screening which, in the opinion of the investigator, could affect the natural course of the disease and thus affect the evaluation of the treatment.
* History of any active skin infection within 1 week prior to baseline.
* Clinically significant infection within 4 weeks prior to baseline which, in the opinion of the investigator, could compromise the safety of the subject in the trial, interfere with evaluation of the IMP, or reduce the subject's ability to participate in the trial. Clinically significant infections are defined as:

  * A systemic infection.
  * A serious skin infection requiring parenteral (intravenous or intramuscular) antibiotics, antiviral, or antifungal medication.
* Tuberculosis requiring treatment within 12 months prior to screening and/or subjects with a positive blood test for tuberculosis at screening. Subjects with high risk of latent tuberculosis (e.g. prior residence in or travel to countries with high prevalence of tuberculosis, close contact with a person with active tuberculosis, or a history of active or latent tuberculosis where an adequate course of treatment cannot be confirmed) must have been tested at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (19):
- United States (5):
  - LEO Pharma Investigational Site, San Diego, California
  - LEO Pharma Investigational Site, Skokie, Illinois
  - LEO Pharma Investigational Site, Boston, Massachusetts
  - LEO Pharma Investigational Site, Forest Hills, New York
  - LEO Pharma Investigational Site, Cincinnati, Ohio
- Denmark (3):
  - LEO Pharma Investigational Site, Aarhus
  - LEO Pharma Investigational site, Hellerup
  - LEO Pharma Investigational Site, Odense
- France (4):
  - LEO Pharma Investigational Site, Loiré
  - LEO Pharma Investigational Site, Nice
  - LEO Pharma Investigational Site, Paris
  - LEO Pharma Investigational Site, Toulouse
- Germany (7):
  - LEO Pharma Investigational Site, Aachen
  - LEO Pharma Investigational Site, Berlin
  - LEO Pharma Investigational Site, Bochum
  - LEO Pharma Investigational Site, Dresden
  - LEO Pharma Investigational Site, Düsseldorf
  - LEO Pharma Investigational Site, Erlangen
  - LEO Pharma Investigational Site, Oldenburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 subjects screened. 27 subjects randomised. 26 subjects completed.
Pre-assignment Details: A screening visit took place 7 to 28 days before the first application of investigational medicinal product (IMP). To be eligible for participation in the trial each subject had to have at least 2 discoid lupus erythematosus (DLE) target lesions with active disease (referred to as lesions 1 and 2) fulfilling the inclusion criteria.
Groups:
- All Subjects: All 27 subjects received delgocitinib cream 20 mg/g on one DLE target lesion and delgocitinib cream vehicle on another DLE target lesion twice daily for 6 weeks.
  Delgocitinib cream 20 mg/g: Cream for topical application.
  Delgocitinib cream vehicle: The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
Period: Overall Study
Arm/Group | All Subjects
Started | 27
Lesions Treated With Delgocitinib Cream (All subjects had one target lesion treated with delgocitinib cream) | 27
Lesions Treated With Delgocitinib Cream Vehicle (All subjects had one target lesion treated with delgocitinib cream vehicle) | 27
Completed | 26
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Randomised subjects
Groups:
- All Randomised Subjects: Randomised subjects received delgocitinib cream 20 mg/g on one DLE target lesion and delgocitinib cream vehicle on another DLE target lesion twice daily for 6 weeks.
  Delgocitinib cream 20 mg/g: Cream for topical application.
  Delgocitinib cream vehicle: The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
Arm/Group | All Randomised Subjects
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 2
  Race: White | 20
  Race: Other | 4
  Race: Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4
  Denmark | 1
  France | 5
  Germany | 17
Investigator's Global Assessment (IGA) of lesions to be treated with delgocitinib cream [Number; unit: percentage of lesions] — The IGA is an instrument used in clinical trials to rate the severity of the subject's global disease and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). In this trial, the IGA was a lesion-specific assessment and was evaluated separately for each of the 2 target lesions.
  percentage of lesions
    IGA score 3 (moderate) | 88.9
    IGA score 4 (severe) | 11.1
Investigator's Global Assessment (IGA) of lesions to be treated with vehicle [Number; unit: percentage of lesions] — The IGA is an instrument used in clinical trials to rate the severity of the subject's global disease and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). In this trial, the IGA was a lesion-specific assessment and was evaluated separately for each of the 2 target lesions.
  percentage of lesions
    IGA score 3 (moderate) | 88.9
    IGA score 4 (severe) | 11.1
Baseline erythema score of lesions to be treated with delgocitinib cream [Number; unit: percentage of lesions] — The erythema score is lesion-specific and based on the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) and the Revised CLASI (RCLASI) which are validated scoring systems to assess disease activity and damage in patients with cutaneous lupus erythematosus. The severity of the erythema is scored on a 4-point scale ranging from 0 to 3. The severity is scored from low to high with 0=absent and 3=dark red, purple/violaceous/crusted/haemorrhagic.
  percentage of lesions
    Erythema score 2 | 37.0
    Erythema score 3 | 63.0
Baseline erythema score of lesions to be treated with vehicle [Number; unit: percentage of lesions] — The erythema score is lesion-specific and based on the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) and the Revised CLASI (RCLASI) which are validated scoring systems to assess disease activity and damage in patients with cutaneous lupus erythematosus. The severity of the erythema is scored on a 4-point scale ranging from 0 to 3. The severity is scored from low to high with 0=absent and 3=dark red, purple/violaceous/crusted/haemorrhagic.
  percentage of lesions
    Erythema score 2 | 48.1
    Erythema score 3 | 51.9
Total skin disease activity score of lesions to be treated with delgocitinib cream [Median (Inter-Quartile Range); unit: scores on a scale] — The total skin disease activity score is defined as the sum of the investigator assessed scores for 3 clinical signs (erythema, scaling/hyperkeratosis, oedema/infiltration) of a lesion. Erythema is scored on a 4-point scale from 0 (absent) to 3 (dark red, purple/violaceous/crusted/haemorrhagic), hyperkeratosis/scaling is scored on a 3-point scale from 0 (absent) to 2 (verrucous hyperkeratosis), and oedema/infiltration is scored on a 3-point scale from 0 (absent) to 2 (palpable and visible). The total skin disease activity score ranges from 0 to 7. Higher scores indicate more severe symptoms.
  scores on a scale | 5.0 [4.0 to 6.0]
Total skin disease activity score of lesions to be treated with vehicle [Median (Inter-Quartile Range); unit: scores on a scale] — The total skin disease activity score is defined as the sum of the investigator assessed scores for 3 clinical signs (erythema, scaling/hyperkeratosis, oedema/infiltration) of a lesion. Erythema is scored on a 4-point scale from 0 (absent) to 3 (dark red, purple/violaceous/crusted/haemorrhagic), hyperkeratosis/scaling is scored on a 3-point scale from 0 (absent) to 2 (verrucous hyperkeratosis), and oedema/infiltration is scored on a 3-point scale from 0 (absent) to 2 (palpable and visible). The total skin disease activity score ranges from 0 to 7. Higher scores indicate more severe symptoms.
  scores on a scale | 5.0 [4.0 to 6.0]

OUTCOME MEASURES:

1. Primary Outcome: Target Lesions With Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 6.
Description: The IGA is an instrument used in clinical trials to rate the severity of the subject's global disease and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). In this trial, the IGA was a lesion-specific assessment and was evaluated separately for each of the 2 target lesions.
Time Frame: Week 6
Population: Per protocol (PP) analysis set. 5 subjects were excluded from the per protocol (PP) analysis set as the primary endpoint data were compromised. The PP analysis set hence comprised 22 (81.5%) subjects. Data at Week 8 was excluded from the PP analysis set for 2 subjects, as they used prohibited concomitant medication in the safety follow-up period.
Measure: Number; unit: lesions
Arm/Group | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 22 | 22
lesions | 3 | 6
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; Test type: Superiority; p = 0.4531, McNemar — Exact p-value of McNemar's test; Attributable risk = -0.14, 95% CI 2-sided [-0.37 to 0.09] — Attributable risk is defined as the difference in estimated probability of treatment success of delgocitinib compared to vehicle. Exact p-value of McNemar's test. Success is defined as having an IGA score of 0 (clear) or 1 (almost clear) at Week 6

2. Secondary Outcome: Number of Adverse Events (AEs) up to Week 6.
Description: Number of AEs from baseline to Week 6
Time Frame: Week 0 to Week 6
Population: Safety analysis set. All 27 subjects were exposed to IMP. All subjects were treated with delgocitinib cream on one target lesion and with vehicle on another target lesion, and except for lesion-specific AEs, it was therefore not possible to distinguish between AEs related to delgocitinib cream or vehicle treatment.
Measure: Number; unit: AEs
Groups:
- All Subjects: All subjects received delgocitinib cream 20 mg/g on one DLE target lesion and delgocitinib cream vehicle on another DLE target lesion twice daily for 6 weeks.
  Delgocitinib cream 20 mg/g: Cream for topical application.
  Delgocitinib cream vehicle: The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
Arm/Group | All Subjects
Number analyzed (Participants) | 27
AEs | 8

3. Secondary Outcome: Number of Subjects With AEs up to Week 6.
Description: Number of subjects with AEs from baseline to Week 6
Time Frame: Week 0 to Week 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 27
Participants | 8

4. Secondary Outcome: Number of Lesion-specific, Treatment-related AEs up to Week 6.
Description: The number of lesion-specific, treatment-related AEs per target lesion will be compared for active and vehicle treatment. Lesion-specific AEs are defined as lesional/perilesional AEs (i.e. AE location within the treatment area and/or ≤2 cm from the border of a target lesion).
Time Frame: Week 0 to Week 6
Population: Safety analysis set. All 27 subjects were exposed to IMP. All subjects were treated with delgocitinib cream on one target lesion and with vehicle on another target lesion. It was therefore only possible to distinguish between AEs related to delgocitinib cream or vehicle treatment for the lesion-specific AEs.
Measure: Number; unit: AEs
Arm/Group | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 27 | 27
AEs | 2 | 0
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; Test type: Superiority; p = 0.5000, McNemar — Exact p-value of McNemar's test; Attributable risk = 0.07, 95% CI 2-sided [-0.02 to 0.17] — Attributable risk is defined as the difference in estimated probability of treatment success (i.e. no lesion-specific treatment-related AEs) of delgocitinib compared to vehicle. Exact p-value of McNemar's test

5. Secondary Outcome: Number of Lesions With ≥2-point Reduction in IGA Score at Week 6 Compared to Baseline.
Description: as for outcome 1
Time Frame: Week 0 to Week 6
Population: as for outcome 1
Measure: Number; unit: lesions
Arm/Group | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 22 | 22
lesions | 3 | 6
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; Test type: Superiority; p = 0.4531, McNemar — Exact p-value of McNemar's test; Attributable risk = -0.14, 95% CI 2-sided [-0.37 to 0.09] — Attributable risk is defined as the difference in estimated probability of treatment success of delgocitinib vs vehicle. Exact p-value of McNemar's test. Success is defined as having at least a 2-point reduction in IGA score from baseline to Week 6

6. Secondary Outcome: Number of Lesions With ≥2-point Reduction in Erythema Score at Week 6 Compared to Baseline.
Description: The erythema score is lesion-specific and based on the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) and the Revised CLASI (RCLASI) which are validated scoring systems to assess disease activity and damage in patients with cutaneous lupus erythematosus. The severity of the erythema is scored on a 4-point scale ranging from 0 to 3. The severity is scored from low to high with 0=absent and 3=dark red, purple/violaceous/crusted/haemorrhagic.
Time Frame: Week 0 to Week 6
Population: as for outcome 1
Measure: Number; unit: lesions
Arm/Group | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 22 | 22
lesions | 5 | 5
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; Test type: Superiority; p = 1.0000, McNemar — Exact p-value of McNemar's test; Attributable risk = 0.00, 95% CI 2-sided [-0.22 to 0.22]; Attributable risk is defined as the difference in estimated probability of treatment success of delgocitinib compared to vehicle. Exact p-value of McNemar's test. Success is defined as having at least a 2-point reduction in IGA score from baseline to Week 6

7. Secondary Outcome: Erythema Score at Week 6.
Description: The erythema score is lesion-specific and based on the CLASI and the RCLASI which are validated scoring systems to assess disease activity and damage in patients with cutaneous lupus erythematosus. The severity of the erythema is scored on a 4-point scale ranging from 0 to 3. The severity is scored from low to high with 0=absent and 3=dark red, purple/violaceous/crusted/haemorrhagic.
Time Frame: Week 6
Population: Per protocol (PP) analysis set.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 22 | 22
scores on a scale | 1.5 [1 to 2] | 1.5 [1 to 2]
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; Test type: Superiority; p = 0.5797, Wilcoxon signed rank test — P-value of the Wilcoxon signed rank test; Erythema is scored as 0=absent, 1=pink, faint, 2=red, 3=dark red, purple/violaceous/crusted/haemorrhagic. P-value of the Wilcoxon signed rank test

8. Secondary Outcome: Total Skin Disease Activity Score (Sum of Scores for Erythema, Scaling/Hyperkeratosis, and Oedema/Infiltration) at Week 6.
Description: The skin disease activity scores are based on the CLASI and the RCLASI which are validated scoring systems to assess disease activity and damage in patients with cutaneous lupus erythematosus. The total skin disease activity score is defined as the sum of the scores for 3 clinical signs (erythema, scaling/hyperkeratosis, oedema/infiltration) for each target lesion. For the total score and the individual clinical signs, higher scores indicate more severe symptoms. Erythema is scored on a 4-point scale ranging from 0 (absent) to 3 (dark red, purple/violaceous/crusted/haemorrhagic). Hyperkeratosis/scaling is scored on a 3-point scale from 0 (absent) to 2 (verrucous hyperkeratosis). Oedema/infiltration is scored on a 3-point scale from 0 (absent) to 2 (palpable and visible). The total skin disease activity score can therefore range from 0 to 7.
Time Frame: Week 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 22 | 22
scores on a scale | 2.5 [2 to 4] | 2.5 [1 to 4]
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; Total skin disease activity score is the sum of the scores for erythema, scaling/hyperkeratosis, and oedema/infiltration. Total skin disease activity score ranges from 0 to 7 with lower score indicating better state; Test type: Superiority; p = 0.7862, Wilcoxon signed rank test — P-value of the Wilcoxon signed rank test; P-value of the Wilcoxon signed rank test

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: All 27 subjects in the safety analysis set were treated with delgocitinib cream on one target lesion and with vehicle on another target lesion, and except for lesion-specific AEs, it was therefore not possible to distinguish between AEs related to delgocitinib cream or vehicle treatment.
Groups:
- All Subjects: All 27 subjects in the safety analysis set were treated with delgocitinib cream on one target lesion and with vehicle on another target lesion, and except for lesion-specific AEs, it was therefore not possible to distinguish between AEs related to delgocitinib cream or vehicle treatment.
  Delgocitinib cream 20 mg/g: Cream for topical application.
  Delgocitinib cream vehicle: The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 10/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=27)
Nasopharyngitis (Infections and infestations) | 4 (5)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 (1) — This lesion-specific AE was assessed as probably related to delgocitinib cream, and the lesion was recovered/resolved from this AE. The subject was withdrawn from the trial due to this AE.
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Application site pain (General disorders) | 1 (2) — This lesion-specific AE was assessed as possibly related to delgocitinib cream, and the lesion was recovered/resolved from this AE.
Application site pruritus (General disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated prematurely due to slow recruitment, and due to an anticipation that recruitment would become further delayed due to the COVID-19 pandemic affecting recruitment activities. The total number of subjects included in the trial therefore ended with 27 subjects randomised. 26 subjects completed the trial, as 1 subject withdrew from the trial due to an AE (moderate cutaneous lupus erythematosus [CLE]; reported term: cutaneous lupus erythematosus flare).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma A/S seeks publication of all clinical trials in peer-reviewed journals within 18 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by LEO Pharma A/S within these 18 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03958955/Prot_SAP_000.pdf